CLINICAL TRIAL: NCT05732311
Title: Intermittent Theta Burst Stimulation for Maintenance Therapy in Depression
Acronym: PROTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Berthold Langguth, MD, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Berthold Langguth, MD, Ph.D., Prof. Dr., University of Regensburg
Organization: University of Regensburg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-3167-101
Record Dates: First submitted 2023-02-07; First posted 2023-02-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active treatment (Experimental): 600 pulses of iTBS per day with 120% resting motor threshold applied five days in one week; tapering interval over 8 months (three treatments with breaks of three weeks; two treatments with breaks of five weeks; one last treatment after eight weeks)
  Interventions: Device: intermittend theta burst stimulation
- active treatment 2 (Active Comparator): 600 pulses of iTBS per day with 120% resting motor threshold applied five sessions in one day (three treatments with breaks of three weeks; two treatments with breaks of five weeks; one last treatment after eight weeks)
  Interventions: Device: intermittend theta burst stimulation

INTERVENTIONS:
Device: intermittend theta burst stimulation — intermittend theta burst stimulation

SUMMARY:
This is a randomized, multi-center, open-label study in which patients with depression who responded to an open-label treatment with intermittent theta burst stimulation (iTBS) will receive this procedure as maintenance therapy. The patients will be randomized to two study arms. The arms differ in the frequency of stimulation (standard iTBS (5 treatments every working day for one week) vs. accelerated iTBS (5 treatments in one day)). For purposes of effect size estimation an interim analysis will be done after half of the patients.

ELIGIBILITY:
Inclusion Criteria:

* adult women and men aged 18 to 70 years with an ICD-10 diagnosis of a depressive episode of depressive disorder (F32), recurrent depressive disorder (F33), or bipolar disorder (F31)
* moderate or severe current episode prior to initial open iTBS treatment (HAMD-21 >16 points)
* response to iTBS treatment (either reduction in HAMD score by 50% or score at the end of treatment <11 points)
* no concomitant psychotic symptoms.
* no other relevant psychiatric disorder as assessed by the study physician
* residence in Germany and German speaking that allows understanding of the information provided
* patient is capable of giving consent

Exclusion Criteria:

* fulfillment of the general contraindications for TMS (electrical implants or metallic objects in the body such as pacemakers or insulin pumps).
* severe neurological diseases (e.g., cerebrovascular events, neurodegenerative diseases, epilepsy, malformations of the brain, severe head injury in the history)
* current harmful use or dependence on alcohol, amphetamines, cocaine, benzodiazepines, anticonvulsants, or opiates
* acute suicidality
* pregnancy
* current participation in another study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
relapse (number of patients who have a relapse for depression) | 33 weeks
  50% increase of symptoms according to Hamilton depression rating scale

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | 49 weeks
  Hamilton Depression Rating Scale (range: 0-65; higher values = worse outcome)
Major Depression Inventory | 49 weeks
  Major Depression Inventory (range: 0-50; higher values = worse outcome)
World Health Organisation quality of life bref | 49 weeks
  World Health Organisation quality of life bref (range: 4-20; lower values = worse outcome)
clinical global impression | 49 weeks
  clinical global impression (range: 0-7; higher values = worse outcome)
Columbia-Suicide Severity Rating Scale | 49 weeks
  Columbia-Suicide Severity Rating Scale (range: 0-6; higher values = worse outcome)
Beck Anxiety Index | 49 weeks
  Beck Anxiety Index (range: 0-63; higher values = worse outcome)
Global Assessment of Functioning | 49 weeks
  Global Assessment of Functioning (range: 0-100; lower values = worse outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, Prof., Principal Investigator — University Hospital of Regensburg, Department of Psychiatry and Psychotherapy at the Bezirksklinikum
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No